CLINICAL TRIAL: NCT07217535
Title: The Rutgers University Study of the Genetics of Kidney Disease
Brief Title: Rutgers University Study of the Genetics of Kidney Disease
Acronym: rugcc-kd
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Tara Matise, Ph.D., Distinguished Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2025001024
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Kidney Disease; Kidney Disease, Chronic; Kidney Disease, End-Stage; Kidney Diseases; Kidney Diseases, Chronic; Kidney Diseases,Cystic
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Kidney Diseases, Cystic | interventions — Health Surveys

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney disease cases: Study participants who have been diagnosed with any form of kidney disease, either currently or in the past.
  Interventions: Genetic: Saliva sample; Other: Health surveys
- Kidney disease controls: Study participants who have never been diagnosed with any form of kidney disease, either currently or in the past.
  Interventions: Genetic: Saliva sample; Other: Health surveys

INTERVENTIONS:
Genetic: Saliva sample — Saliva sample is sent via prepaid US Mail for DNA extraction
Other: Health surveys — Health surveys are filled out online in the study portal.

SUMMARY:
The goal of this observational study is to learn more about how genes impact the risk of kidney disease. Anyone 18 or older living in the US is eligible, and a diagnosis of kidney disease is NOT required. Study participation is online, and it takes about 20 minutes to complete health surveys and request a saliva collection kit sent through US mail. In return, study participants may opt to receive information about their genetic ancestry at no cost.

DETAILED DESCRIPTION:
This is an online research study to learn more about how genes affect the risk of kidney disease. This is an online research study to learn more about how genes affect the risk of kidney disease. No office visit is required and in return, participants may receive information about their genetic ancestry for free. One in seven individuals in the United States today has chronic kidney disease (CDC 2023). The heritability -a measure of genetic, as opposed to environmental, contribution to a disease- of kidney function such as the estimated glomerular filtration rate (eGFR) has been estimated at 38%This study will increase our understanding of the genetic basis of kidney disease, which is a crucial step in drug development to improve current treatment options. The study investigators seek a diverse population because diversity among participants maximizes the usefulness of the data. Participants will use our online study portal to answer questions about their health and provide their DNA via a saliva sample using a pre-paid mailer. Participation takes approximately 20 minutes. Participants will be invited to share data from their electronic health records, but this is not required for study participation. The study investigators keep participants engaged with short monthly newsletters.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* currently living in the United States
* able to understand and follow written instructions in English
* have access to the internet and a computer, laptop, tablet or smart phone
* willing to provide written informed consent for participation
* willing to provide DNA via a saliva sample using a collection kit mailed to the study participant's home
* willing to complete a survey with questions about health related to the study of kidney disease

Exclusion Criteria:

* Not able to meet or fulfill any of the inclusion criter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of anyone at least 18 years old who lives in the United States, including both individuals who have or had kidney disease and those who have not. Participants include males, females, non-binary, and all race-ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Genetic risk variants associated with kidney disease | 2 years
  Genetic factors will be measured through whole exome sequencing along with genotyping of common variants, and then correlated with kidney disease and/or kidney disease subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Matise, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, The State University of New Jersey, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website with information about the study — https://rugcc.rutgers.edu/kidney-disease/